CLINICAL TRIAL: NCT06143800
Title: The Effect and Underlying Mechanism of Reconsolidation-Based Cognitive Reappraisal for Traumatic Memories in Patients With Major Depression Disorder
Brief Title: Reconsolidation-Based Intervention for Traumatic Memories
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Kangning Hospital (Other)
Collaborators: Science and Technology Innovation Commission of Shenzhen Municipality (Other)
Responsible Party: Principal Investigator, Jingchu Hu, Principal Investigator, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JCYJ20220530165003007
Record Dates: First submitted 2023-10-31; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Psychological Trauma; Memory
MeSH Terms: conditions — Depression; Psychological Trauma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- retrieval + self-focused cognitive reappraisal (Experimental): Participants in this arm will first accept a memory reactivation to open the reconsolidation window, then accept the self-focused cognitive reappraisal intervention.
  Interventions: Behavioral: reactivation; Behavioral: cognitive reappraisal intervention
- retrieval + context-focused cognitive reappraisal (Experimental): Participants in this arm will first accept a memory reactivation to open the reconsolidation window, then accept the context-focused cognitive reappraisal.
  Interventions: Behavioral: reactivation; Behavioral: cognitive reappraisal intervention
- non-retrieval + self-focused cognitive reappraisal (Active Comparator): Participants in this arm will directly accept the self-focused cognitive reappraisal intervention without memory reactivation.
  Interventions: Behavioral: cognitive reappraisal intervention
- non-retrieval + context-focused cognitive reappraisal (Active Comparator): Participants in this arm will directly accept the context-focused cognitive reappraisal intervention without memory reactivation.
  Interventions: Behavioral: cognitive reappraisal intervention

INTERVENTIONS:
Behavioral: reactivation — During the retrieval phase, cues are presented to participants to reactivate their memories; participants in the non-retrieval group go directly to cognitive reappraisal phase.
  Other Names: memory retrieval
  Arms: retrieval + context-focused cognitive reappraisal; retrieval + self-focused cognitive reappraisal
Behavioral: cognitive reappraisal intervention — Subsequently, in the self-focused cognitive reappraisal group, participants will be instructed to use "disengagement" reappraisal to separate themselves from the picture situation and draw a subjective distance so as not to strongly feel the negative emotions brought by the picture. In the context-focused reappraisal group, participants will focus on the picture situation, reappraise the meaning of the picture situation, and assign positive meanings to it.

SUMMARY:
The goal of this clinical trial is to test the effect and underlying mechanism of reconsolidation-based cognitive reappraisal for traumatic memories in patients with major depression disorder. The main questions it aims to answer are:

* Is cognitive reappraisal based on memory reconsolidation effective for laboratory-created traumatic memories? Which of the two classical cognitive reassessment schemes is more effective?
* What is the neural mechanism by which the novel cognitive reappraisal based on memory reconsolidation alters traumatic memories?
* Can repeated use of the novel cognitive reappraisal based on memory reconsolidation alter the actual childhood traumatic memories of patients with major depression disorder? Can it reduce depressive symptoms? Are the effects long-lasting? Participants will be grouped to receive the intervention (retrieval + cognitive reappraisal, non-retrieval + cognitive reappraisal). The researchers will compare the differences in long-term memory tests and the improvement in depressive symptoms between the two groups to see the effects of the memory-based reconsolidation intervention.

DETAILED DESCRIPTION:
There are three sub-trials in this study. Participants in the first trial will learn the fear of emotional faces based on the Pavlovian conditioned fear learning paradigm. Using an inter-subject experimental design, the intervention will be divided into four groups (retrieval /non-retrieval, self-concerned cognitive reappraisal/context-concerned cognitive reappraisal). The researchers will compare the differences between the four groups on long-term memory tests to see if the cognitive reappraisal based on memory reconsolidation has effect on traumatic memory in the laboratory of depressed patients.

Participants in the second trial are given the same treatment as in the first, but with brain imaging equipment to gain brain imaging data. The researchers will compare the brain functional characteristics of the four groups in the long-term memory test, in order to explore the neural mechanism of the effect of cognitive reappraisal on traumatic memory intervention based on memory reconsolidation mechanism.

Participants in the third trial are divided into two groups (retrieval + cognitive reappraisal, and non-retrieval + cognitive reappraisal) for an eight-week intervention. Finally, the researchers will compare the improvement in depressive symptoms between the two groups and retest physiological arousal and subjective assessments of traumatic memories one year later to see the long-term effects of the memory-based reconsolidation intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depression disorder
* Must have normal vision or corrected vision

Exclusion Criteria:

* Have physical diseases or other mental disorders
* Be pregnant, breastfeeding or do not have menstruation
* Drink alcohol or smoke within 24 hours before the experiment
* Participated in similar experiments before.
* History of severe cardiovascular and cerebrovascular diseases, stroke and other neurological diseases, and history of digestive system diseases.
* Severe hearing and vision impairment.
* Have metal implants in the body, such as non-removable dentures, scaffolds, steel plates, joint metal replacements, etc.
* Have Claustrophobia
* Have acute or chronic disease or infection

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Participants' Skin Conductance Response (SCR) | baseline, 8 weeks, and one year after treatment
  The level of SCR was assessed for each trial as the base-to-peak amplitudedifference in skin conductance of the largest deflection (in microsiemens; pS) in the 0.5-4.5-slatency window after stimulus onset.
Change in the amygdala measured with fMRI | baseline, 8 weeks, and one year after treatment
  Changes in the difference in BOLD (Blood Oxygenation Level Dependent) signal in the amygdala between treated cue and untreated cue measured with fMRI.
Change in the hippocampus measured with fMRI | baseline, 8 weeks, and one year after treatment
  Changes in the difference in BOLD (Blood Oxygenation Level Dependent) signal in the hippocampus between treated cue and untreated cue measured with fMRI.
Change in the prefrontal cortex measured with fMRI | baseline, 8 weeks, and one year after treatment
  Changes in the difference in BOLD (Blood Oxygenation Level Dependent) signal in the prefrontal cortex between treated cue and untreated cue measured with fMRI

SECONDARY OUTCOMES:
The changes in the Baker Depression Scale (BDI). | baseline, 8 weeks, and one year after treatment
  To assess depressive symptom changes after the treatment using the Baker Depression Scale (BDI). The BDI consists of 21 items coded on a 4-point scale (0-3). The total scores ranged from 0 to 63. The higher the total scores, the higher the depressive symptom severity.
The changes in the State-Trait Anxiety Scale (STAI) | baseline, 8 weeks, and one year after treatment
  To assess anxious symptom changes after the treatment using the State-Trait Anxiety Scale (STAI). The STAI consists of 40 items. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
The changes in the GROSS Self-Rating Emotional Regulation Style Questionnaire | baseline, 8 weeks, and one year after treatment
  To assess emotional regulation style changes after the treatment using the GROSS Self-Rating Emotional Regulation Style Questionnaire. It is a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) Cognitive Reappraisal and (2) Expressive Suppression. Respondents answer each item on a 7-point Likert-type scale (1 to 7). Items 1, 3, 5, 7, 8, 10 make up the Cognitive Reappraisal facet. Items 2, 4, 6, 9 make up the Expressive Suppression facet. Scoring is kept continuous. Each facet's scoring is kept separate.

CONTACTS AND LOCATIONS:
Overall Officials: Jingchu Hu, Dr., Principal Investigator — Shenzhen Kangning Hospital

IPD SHARING:
Plan to Share IPD: Yes
We wiil share our data on the Open Science Framework after data collection
Supporting Information: Study Protocol, SAP
Time Frame: These information will be shared after the related paper is published and will be available for at least one year
Access Criteria: The information will be shared on the Open Science Framework for the public